CLINICAL TRIAL: NCT00973427
Title: DNA Chip Based Prognosis of Lung Cancer
Status: Completed | Type: Observational
Sponsor: Medical Prognosis Institute A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: MPI-1001; H-B-2007-099; WIRB Protocol #20080904
Record Dates: First submitted 2009-09-08; First posted 2009-09-09 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — post resection specimen
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to determine whether a DNA chip, designed by Medical Prognosis Institute (MPI), can provide an accurate prognosis for survival of NSCLC (adeno-, squamous and large cell lung cancer).

ELIGIBILITY:
Inclusion Criteria:

1. A histological diagnosis of primary NSCLC stage Ia
2. Surgical removal of the tumor
3. Age between 18 and 75 years
4. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. A primary NSCLC stage Ia diagnosis that is changed to not primary NSCLC or NSCLC stage Ib-IV after surgery.
2. Adjuvant treatment with chemotherapy.
3. Prior history of cancer in the past 5 years or breast cancer at any time.
4. Life expectancy less than 3 years in the opinion of the investigator due to concurrent illnesses.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population consist of subjects being examined for NSCLC at Roswell Park Cancer Institute (US), University of Alabama (US), Copenhagen University (DK), Odense University Hospital (DK) and Aarhus University Hospital (DK)
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2008-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Disease-related survival | 5 years

SECONDARY OUTCOMES:
Time to progression | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Steen Knudsen, PhD, Study Chair — Medical Prognosis Institute (MPI); Jens B. Sørensen, MD, Study Director — Dept. Oncology, Copenhagen University; Jesper Ravn, MD, Study Director — University of Copenhagen
Locations (5):
- United States (2):
  - University of Alabama, Birmingham, Alabama
  - Roswell Park Cancer Institute, Buffalo, New York
- Denmark (3):
  - Aarhus University Hospital, Aarhus
  - University of Copenhagen, Copenhagen
  - Odense University Hospital, Odense